CLINICAL TRIAL: NCT05099939
Title: Identification of Dysglycemia With Continuous Glucose Monitoring: A Prospective Study to Assess the Relationship With Clinical Evolution in Cystic Fibrosis
Brief Title: Identification of Dysglycemia With Continuous Glucose Monitoring to Assess Clinical Evolution in Cystic Fibrosis
Acronym: ProspeC-F
Status: Recruiting | Type: Observational
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other); University Hospital, Strasbourg, France (Other); Centre Hospitalier Lyon Sud (Other); Fondation Francophone pour la Recherche sur le Diabete (Other)
Responsible Party: Sponsor
Other Study IDs: ProspeC-F
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
Keywords: Diabetes; Screening Test; Continuous glucose monitoring; Oral glucose tolerance test
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cystic fibrosis (CF)-related diabetes (CFRD) is the most important emerging complication after pulmonary complications. This specific form of diabetes is associated with an increased morbidity and mortality. CFRD prevalence at the age of 10 is 10% and reaches 40 to 50% in adulthood, while a similar percentage is afflicted with milder dysglycemia also called pre-diabetes abnormalities.

In order to identify patients at risk and to implement early therapeutic measures, an annual CFRD screening test is recommended for CF patients after 10 years of age. The standard 2-hour oral glucose tolerance test (OGTT) is the recommended screening test. However, this test is perceived by both patients and CF care teams as unpleasant while adding a significant burden and workload, resulting in screening rates lower than 50% in most centers. An ideal alternative test should be simpler, less invasive, more sensitive than an OGTT to establish risks for lung function and/or nutritional deterioration, and predict future CFRD risk. To date, compared to the OGTT, no alternative screening method has demonstrated its effectiveness. However, continuous glucose monitoring (CGM) is emerging as a possible alternative method.

In patients living with CF, CGM is easy to use and can identify early dysglycemia, which in turn, can predict increased risk of accelerated decline of pulmonary function and/or weight, higher risk of pseudomonas colonization, and future risk of CFRD. However, these observations are based on studies of small sample size with very limited prospective data. Furthermore, many of the multiple CGM metrics that have been standardized are based on the risk of complications associated with Type 1 and Type 2 Diabetes.

Thus, there is a need for prospective studies to identify the CGM metrics and the cut-off level that is relevant as a predictor of clinical deterioration and/or CFRD risk in CF. The identification of such CF-specific criteria would provide important information to target at-risk patients.

DETAILED DESCRIPTION:
The investigators propose an international multicenter observational study to evaluate the predictive value of CGM variables on the evolution of the clinical state in adult patients with CF.

To do this, the following will be evaluated:

* The clinical condition of the patients over a period of 5 years (2 years before, up to 3 years after inclusion);
* The detailed glycemic profile using a CGM system during 3 visits (on inclusion, 1 year, then 2 years after inclusion).

The primary objective is to identify which CGM variable, at inclusion in the study, is the most strongly linked to the risk of a decrease in pulmonary function of more than 2% / year measured by the FEV1% over the 5 years of follow-up of the study. The investigators will also i) investigate which CGM variables are most strongly linked to other clinical markers (ex. nutritional status, CFRD diagnosis and pulmonary exacerbations; ii) assess the association between changes in CGM variables (ex. increased number of glycemic excursions >11.0 mmol/L over 2 years) and changes in clinical status over time; and iii) evaluate the correlation between plasma glucose values during the standard routine OGTT and CGM values.

This study includes 3 visits with participants: inclusion (V1), the visit at 1 year (V2), then 2 years after inclusion (V3).

This study consists of 3 phases:

* Phase 1: A retrospective file-based data collection, which covers 2 years before inclusion;
* Phase 2: Prospective data collection, including the installation of a CMG 3 times over a period of 2 years, then;
* Phase 3: An additional one-year prospective data collection on file only.

Only phase 2 includes visits for the participant. A CMG system will be installed for 14 days at inclusion (visit 1), at 1 year (visit 2) and 2 years (visit 3) during a regular routine visit and / or an annual OGTT visit. The participants' only involvement will be to wear the CMG system and return it to the research center at the end of the 14-day period. All data obtained during a routine visit will be collected directly from medical records over a period of 5 years (two years before inclusion until the final visit): pulmonary function (FEV1), nutritional status (weight and height), bronchial colonization by Pseudomonas aeruginosa, number of exacerbations, number of intravenous antibiotic courses, number of hospitalizations, and annual OGTT results.

ELIGIBILITY:
Inclusion Criteria:

* Have cystic fibrosis
* Be 18 years of age or older
* Have given clear and informed consent

Exclusion Criteria:

* Receive pharmaceutical treatment for diabetes
* Have had a lung or liver transplant
* Participate in a randomized controlled trial for more than 3 months in parallel with this study
* Currently pregnant
* Patients under legal protection (for centers in France)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals living with cystic fibrosis who are being followed at the following centers: Centre Hospitalier de l'Université de Montréal (CHUM), Université de Lyon (Hospices Civils de Lyon) and Université de Strasbourg (CHU de Strasbourg).
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in lung function | 5 years
  The primary outcome is the mean annual rate of change in lung function (FEV1%) from 2 years before inclusion to 3 years later, for a total of 5 years of follow-up.

SECONDARY OUTCOMES:
Change in body mass index | 2 years
  Change in body mass index weight category from inclusion to 2 years (underweight, adequate weight, overweight).
Number of pulmonary exacerbations | 1 year
  Average annual number of pulmonary exacerbations per year (validated Fuchs questionnaire), including exacerbations that are treated at home or at the hospital.
CFRD diagnosis | 3 years
  Development of new cases of CFRD diagnosed with standard OGTT and initiation of all anti-diabetic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal; Laurence Kessler, Principal Investigator — CHU de Strasbourg; Isabelle Durieu, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- Canada (2):
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
- France (2):
  - Hospices Civils de Lyon, Lyon
  - CHU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No